CLINICAL TRIAL: NCT02941497
Title: "Get Fruved:" A Peer-led, Train-the-trainer Social Marketing Intervention to Increase Fruit and Vegetable Intake and Prevent Childhood Obesity.
Brief Title: Get Fruved: Obesity Prevention for Older Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Florida (Other); West Virginia University (Other); South Dakota State University (Other); Auburn University (Other); Syracuse University (Other); University of Maine (Other); Kansas State University (Other)
Responsible Party: Principal Investigator, Sarah Colby, Associate Professor, The University of Tennessee, Knoxville
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UTK IRB-14-09366 B-XP; 2014-67001-21851 (Other Grant/Funding Number: USDA National Institute of Food and Agriculture A2101); WBS number R011770127 (Other: University of Tennessee)
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Stress, Psychological; Obesity; Physical Activity; Fruit; Vegetables; Social Marketing; Peer Influence; Community-Based Participatory Research
MeSH Terms: conditions — Obesity; Stress, Psychological; Motor Activity | interventions — Social Marketing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive intervention group (Experimental): The intensive intervention group participates in development and implementation of the social marketing and health promotion campaign and peer-led campus activities and is assessed for their health-related behaviors. This was Wave 1 in colleges in Yr 01-02 and is being repeated as Wave 2 in colleges in Yr 03. This will also be repeated in high schools in Yr 04.
  Interventions: Behavioral: Social marketing and health promotion campaign
- Diffuse intervention group (Experimental): The diffuse intervention group receives the social marketing and health promotion campaign and participates in the peer-led campus activities and is assessed for their health related behaviors, but is not involved in the design and delivery of the intervention materials and activities. This was Wave 1 in colleges in Yr 01-02 and is being repeated as Wave 2 in colleges in Yr 03. This will also be repeated in high schools in Yr 04.
  Interventions: Behavioral: Social marketing and health promotion campaign

INTERVENTIONS:
Behavioral: Social marketing and health promotion campaign — Students in the intensive intervention group developed a nine-month social marketing health campaign. The campaign included five costumed characters who interacted with students on campus in residence halls, dining halls, and other highly-trafficked public areas on campus. Photos and videos of interactions were put on social media. Student participants from the general population (the diffuse intervention group) were asked to set weekly healthy goals related to diet, physical activity, and stress management throughout the campaign and received email and text messages with goal-specific written and video health-promotion messages. Faculty partnered with the students throughout the intervention process to educate and give advice on the content of health promotion messages.
  Other Names: Get Fruved

SUMMARY:
This program is a non-diet approach to obesity prevention for older adolescents which does not promote following a special diet to manage weight; it promotes healthy behavior associated with obesity prevention. This approach is important with youth and older adolescent populations to avoid impairment in emotional well-being associated with body dissatisfaction. Healthy weight status will be achieved by improving dietary intake patterns, increasing physical activity, and improving stress management. Fall of year 01 was devoted to the recruitment of student partners (intense intervention group) and the development of partnerships. In the spring of year 01, recruited students were enrolled in two newly developed undergraduate courses across four intervention state partners, became collegiate 4-H members, planned a social marketing campaign, and/or learned to be peer mentors or student researchers. In year 02, first year college students were recruited, peer mentors were matched with a group of first year students, and the developed social marketing campaign was pilot tested on four college campuses (diffuse intervention) by the collegiate 4-H teams. In year 02, a toolkit with 24 weeks of intervention activities was also refined. In year 03, the collegiate 4-H team (intense intervention group) used the refined toolkit to test and implement the intervention on college campuses. In year 03, the assessment process for high school 4-H students (intense intervention group) will be pilot tested and college students will work with the high school students on adapting the toolkit for use in the implementation of the social marketing campaign in high school settings in year 04 (diffuse intervention). ). In year 04, the pilot and feasibility tested college intervention was tested with a randomized control trial design with 30 intervention and 29 control university partners. The adapted high school toolkit was pilot and feasibility tested in three intervention and two control high school settings. In year 05, the high school intervention was tested with a randomized control trial design with 9 intervention and 7 control high schools in one district's high schools. On all measures it is anticipated that participants in the intensive intervention group will have greater improvements than those in the diffuse intervention group and both intensive and diffuse intervention groups will have improvements over those in the control groups.

DETAILED DESCRIPTION:
The goal of the research is to develop a novel strategy to promote healthy behaviors associated with obesity prevention in older adolescent populations. A community based participatory research (CBPR) approach is used with partnerships among older adolescents, university researchers and faculty, and Extension partners. The objective is to test the effectiveness of a peer-led, train-the-trainer intervention. The intervention is an interactive, non-traditional social marketing, online media, and environmental change approach seeking to promote healthy behavior with communities of college and high school students. Specific health behaviors targeted include increasing intakes of fruits and vegetables, decreasing foods high in saturated fats and added sugars, managing stress, and increasing physical activity. This project uniquely 1) increases participant engagement through creative interactions, participant-created content, and incorporation of age-appropriate technology; 2) incorporates social environments and peer-led strategies; and 3) simultaneously addresses changes in environments to support participant-driven behavior change efforts.

This project is a Pretest-Posttest, Control Group Trial using a nested cohort design with three conditions (intense intervention, diffuse intervention, and control), four control universities and four intervention universities in years 01- 03, one high school as control and one as intervention at each of the four intervention university towns in years 03-04, and disseminated to four additional university and high school pairs in years 04-05.

A CBPR, peer-led approach is used in that upper level college students mentor freshmen 4-H college students through the development of the intervention. The CBPR, peer-led approach continues when the now sophomore 4-H college students implement the intervention with incoming college freshmen in the following year. The train-the-trainer approach is utilized when the now junior level 4-H college students mentor 4-H high school students in the modification of the intervention for high schools. The approach continues when 4-H high school students implement the intervention with incoming freshmen in high schools.

In the fall of year 01, 283 freshman students were recruited from general/survey nutrition courses at the four intervention universities to participate in a special undergraduate spring course (the intense intervention group). 94 freshman students were also recruited from general/survey nutrition courses at the four control universities. During the fall, researchers at the intervention schools worked with nutrition (graduate and undergraduate) students to identify and develop partnerships with student organizations for the development of a social marketing health promotion campaign. Researchers and student partners also worked with local high schools (including student organizations, school food service, Parent Teacher Associations, school wellness committees, and administration) and school boards to formalize research agreements and relationships.

In the spring of year 01, as a part of the newly developed undergraduate course, the freshman students (the intense intervention group) from each intervention university joined their collegiate 4-H program. The courses were offered as independent studies or as a newly developed course through the respective University's PI. The course covered principals of social marketing for health behavior change. University researchers and Extension faculty collaborated and taught in-person classes with their respective collegiate 4-H students. Collegiate 4-H students were co-taught (by all four University's research and Extension faculty) and had the opportunity to interact with the other collegiate 4-H students from all four intervention universities through web-based technologies. Throughout the course, the collegiate 4-H students developed and planned a social marketing campaign. Following a peer-led approach, the 4-H students partnered with and were mentored by upper-level nutrition students and student organizations (student partners) in the development and planning of the campaign.

In year 02, the now sophomore collegiate 4-H students in the intense intervention group (receiving hourly compensation) worked with student partners to implement the developed nine-month social marketing campaign. The campaign centered around five costumed characters (Spinach, Carrot, Banana, Grapes, and Tomato). Characters interacted with students on campus in freshmen residence halls, dining halls/cafeterias and highly trafficked public areas on campus. Photos and videos of interactions were put on the website (www.fruved.com), Facebook, twitter, YouTube, Snap Chat, and Instagram. Online educational modules (focused on healthy diet patterns, physical activity, and stress management) will also become available on the website. Student participants from the general freshman population were asked to set weekly healthy goals related to diet, physical activity, and stress management throughout the campaign and receive email and/or text messages with goal-specific written and video health promotion messages. Extension faculty and staff partnered with the collegiate 4-H student teams throughout the intervention process to educate and give advice on the content of health promotion messages. Throughout the campaign, collegiate 4-H students worked with researchers to assess the healthiness of their campus environments using a previously developed Healthy Campus Audit and advocated for changes to the physical and food environment.

In year 02, a random sample of 1,153 freshmen (the diffuse intervention group), determined by screening to be at increased health risk were recruited from the eight universities (four intervention and four control). The collegiate 4-H students (the intense intervention group) and the same students from the control schools recruited in year 01 were reassessed.

In year 03, the collegiate 4-H team (intense intervention group) will use the refined toolkit to test and implement the intervention on college campuses. The sustainability of observed changes at the individual and environmental college level will be assessed by conducting follow-up assessments with the students in the intervention (the diffuse intervention group) and control sites at colleges in year 03. The collegiate 4-H students (the intensive intervention group) leading the project at the high school level and the same students from the control schools recruited in year 01 will be reassessed at the beginning of fall year 03, and end of spring year 03. Also in year 03, the assessment process for high school 4-H students (intense intervention group) will be piloted tested and college students will work with the high school students on adapting the toolkit for use in the implementation of the social marketing campaign in high school settings (diffuse intervention).

In year 04, two high schools in each of the four intervention University states participated in the research process and were randomized to control and intervention. High schools in each state were matched by size and community composition and geographically separated to prevent potential exposure to the campaign. Following the train-the-trainer model, teams of now junior collegiate 4-H students (the intense intervention group) mentored teams of high school 4-H students (the intense intervention group) at each of the intervention sites in the development and implementation of the Fruved campaign in the high school environment. In the fall, collegiate students will work with the high school students (the intense intervention group) to modify the campaign to meet the age and cultural needs of a high school audience and plan the specific campaign components. The high school 4-H teams will partner with their school's food service, Parent Teacher Association (PTA), school Wellness committee, and school administration throughout the campaign development, implementation, and evaluation. The campaign will be conducted in the intervention high schools over the remaining nine-month school year.

In year 04, a random sample of 331 freshman high school students (the diffuse intervention group) will be recruited from the intervention high schools and a random sample of 331 freshman high school students (the control group) from the control high schools in each of the four intervention University town areas. Assessments will take place in early fall and late spring. The 4-H high school students (intensive intervention group) recruited to participate in the design and implementation phases of the project will also be assessed in early fall/late spring in year 04.

Also in year 04, to continue to assess the sustainability of observed changes at the individual and environmental high school level, participants will be assessed by conducting follow-up assessments with the students in the intensive intervention group and control sites in high schools. The collegiate 4-H students (the intensive intervention group) that lead the project at the high school level and the same students from the control schools recruited in year 01 will be reassessed at the beginning of fall year 04 and end of spring year 04.

In year 04-05, materials will be developed allowing the project to be further disseminated to other college and high school environments. Four additional college and high school pairs will be recruited to participate in the dissemination phase. In year 04 the college students will receive training materials, study manual, costumes, cameras, and a small implementation budget but will not receive support for incentives or student 4-H compensation. The campaign will be developed and implemented over one school year. A modified project assessment will be required to be completed by the collegiate student 4H groups. In year 05 the collegiate 4-H students will work with high school 4-H students to develop and implement the project in high schools. The high school 4-H student group will complete the modified project assessments.

The nine month interactive, social marketing environmental intervention will aid older adolescents in effectively preventing obesity through increasing healthfulness of diet, increased physical activity, and improved stress management behavior as compared to a control group. On all measures it is anticipated that participants in the intensive intervention group will have greater improvements than those in the diffuse intervention group and both intensive and diffuse intervention groups will have improvements over those in the control groups. Students participating in the intervention will more effectively manage their weight than those in the non-intervention control condition; those participating in the intervention will improve intermediary outcomes related to diet, physical activity, and improved stress management to a greater extent than those in the control condition; and environments at intervention sites will show health behavior-supportive changes as compared to control sites.

Since there are more than two time intervals in the design, General Linear Modeling will be used to analyze for changes in physical assessments, specifically a mixed-model Analysis of variance and covariance (ANCOVA) if the group-specific slopes are homogeneous. A wide range of analyses will be employed to analyze the influence of the intervention on secondary outcomes, including multivariate analyses of variance (MANOVA), ANOVAs, and logistic regression. Significant ANOVAs will be followed up with tests of simple and main effects as appropriate. The intervention group-by-occasions interaction test will assess the impact of the intervention in the treatment group relative to the control group across time on the secondary outcome measures.

ELIGIBILITY:
Inclusion criteria:

* Students in the intensive intervention group must be registered for a general/survey nutrition or wellness course
* Students in the diffuse intervention group randomly selected from those who screen in because they are at increased health risk (increased BMI and waist circumference, low intakes of fruits and vegetables, high levels of stress, and low levels of physical activity)

Exclusion criteria:

* There are no exclusionary criteria for students in the intensive intervention group
* Students who are not at-risk for health issues are excluded from the diffuse intervention group

Max Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5800 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change in body weight from baseline to six months and one year follow up
  Following an overnight fast and voiding, weight is measured in light clothing without shoes and with pockets emptied. Weight is measured in duplicate (average used unless > 0.1 kg difference requiring re-measurement until 2 values within range are achieved) to the nearest 0.1 kilograms using a calibrated electronic scale by trained assessors. Height without shoes is measured to the nearest 0.1 centimeter using a portable stadiometer. Height and weight are used to calculate BMI.

SECONDARY OUTCOMES:
Amount of physical activity | Change in amount of physical activity from baseline to six months and one year follow up
  The International Physical Activity Questionnaire (IPAQ) is used to measure self-reported physical activity. Results are calculated as Metabolic Equivalent (MET) minutes/week and can be used to estimate energy expenditure.
Dietary quality | Change in dietary quality from baseline to six months and one year follow up
  The Automated Self-Administered Recall System (ASA24) is a web-based tool that allows participants to complete 24-hour recalls online. The Researcher Web site is used to incorporate the recall process in assessments and analyze data. Subjects complete the initial 24-hour recall at the time of the in-person physical assessment. They then receive email prompts asking them to completed two follow-up 24 hour recalls within the same week for a total of two recalls on nonconsecutive weekdays and one weekend day.
Fruit and vegetable intake | Change in fruit and vegetable intake from baseline to six months and one year follow up
  Cups of fruits and vegetables/day is assessed using the NCI Fruit and Vegetable Screener (FVS). The FVS is a 19-item instrument that includes assessment of portion size.
Body composition | Change in body composition from baseline to six months and one year follow up
  All circumference measurements are done using a Gulick tape measure. The waist is measured at the level of the iliac crests. The hips are measured at the maximum extension of the buttocks, and used to calculate body adiposity index (9) and hip to waist ratio. The neck is measured at the level of the Adams apple which can be palpated to identify location.
Eating competence | Change in eating competence from baseline to six months and one year follow up
  Eating competence is measured using ecSatter Inventory (ecSI). The ecSI consists of 16 items that measure eating attitudes, food acceptance, internal regulation, and contextual skills such as meal planning. Those who have higher eating competence scores are more likely to be satisfied with weight, have lower BMI, and consume more fruits and vegetables than those with lower eating competence scores.
Stress | Change in stress from baseline to six months and one year follow up
  Perceived stress is measured Cohen's Perceived Stress Scale (PSS). The PSS is a 14 item instrument designed to measure the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Behavior changeability | Change in perceptions and willingness to change from baseline to six months and one year follow up
  The Behavioral Environmental Changeability Survey (BECS) was developed and is used to assess perceptions of the importance and willingness to change weight related behavior. The BECS consists of eight scales (Nutrition Changeability; Nutrition Behavior; Environmental Changeability; Program Importance and Changeability; Exercise Behavior; Sleep Behavior and Importance; Weight Loss; and Alcohol Intake).
Sleep | Change in sleep from baseline to six months and one year follow up
  Quality and quantity of sleep are assessed using the Pittsburg Sleep Quality Index (PSQI). The survey has 19 self-reported items related to sleep over the past month. The items generate seven component scores (sleep quality, sleep latency, duration, efficiency, disturbances, use of sleeping medication and daytime dysfunction) which are summed for a global PSQI score.
Campus healthy food access | Change in campus food choice from baseline to six months and one year follow up
  Changes in overall consumption of all foods on campus are evaluated by reviewing the ordering records (with control for total student population) and sales data for all vending and dining services.
Environmental change | Change in the campus environment from baseline to six months and one year follow up
  The changes in the environment are assessed using the Healthy Campus Audit and the CEPS. The HCA assesses physical activity, food, and policy aspects of the environment.
Recreational facility usage | Change in recreational facility usage from baseline to six months and one year follow up
  The use of the recreational facilities are assessed through reviewing entrance records (with control for total student population).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Colby, PhD, RD, Principal Investigator — University of Tennessee
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Kansas State University, Manhattan, Kansas
  - University of Maine, Orono, Maine
  - Syracuse University, Syracuse, New York
  - South Dakota State University, Brookings, South Dakota
  - University of Tennessee, Knoxville, Tennessee
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time.

REFERENCES:
- [Background] Byrd-Bredbenner C, Johnson M, Quick VM, Walsh J, Greene GW, Hoerr S, Colby SM, Kattelmann KK, Phillips BW, Kidd T, Horacek TM. Sweet and salty. An assessment of the snacks and beverages sold in vending machines on US post-secondary institution campuses. Appetite. 2012 Jun;58(3):1143-51. doi: 10.1016/j.appet.2012.02.055. Epub 2012 Mar 10. PMID 22414787
- [Background] Do M, Kattelmann K, Boeckner L, Greene G, White A, Hoerr S, Horacek T, Lohse B, Phillips B, Nitzke S. Low-income young adults report increased variety in fruit and vegetable intake after a stage-tailored intervention. Nutr Res. 2008 Aug;28(8):517-22. doi: 10.1016/j.nutres.2008.05.013. PMID 19083454
- [Background] Gordon R, McDermott L, Stead M, Angus K. The effectiveness of social marketing interventions for health improvement: what's the evidence? Public Health. 2006 Dec;120(12):1133-9. doi: 10.1016/j.puhe.2006.10.008. Epub 2006 Nov 13. PMID 17095026
- [Background] Gracia-Marco L, Vicente-Rodriguez G, Borys JM, Le Bodo Y, Pettigrew S, Moreno LA. Contribution of social marketing strategies to community-based obesity prevention programmes in children. Int J Obes (Lond). 2011 Apr;35(4):472-9. doi: 10.1038/ijo.2010.221. Epub 2010 Oct 26. PMID 20975724
- [Background] Greene GW, Schembre SM, White AA, Hoerr SL, Lohse B, Shoff S, Horacek T, Riebe D, Patterson J, Phillips BW, Kattelmann KK, Blissmer B. Identifying clusters of college students at elevated health risk based on eating and exercise behaviors and psychosocial determinants of body weight. J Am Diet Assoc. 2011 Mar;111(3):394-400. doi: 10.1016/j.jada.2010.11.011. PMID 21338738
- [Background] Horacek TM, Erdman MB, Byrd-Bredbenner C, Carey G, Colby SM, Greene GW, Guo W, Kattelmann KK, Olfert M, Walsh J, White AB. Assessment of the dining environment on and near the campuses of fifteen post-secondary institutions. Public Health Nutr. 2013 Jul;16(7):1186-96. doi: 10.1017/S1368980012004454. Epub 2012 Oct 17. PMID 23174458
- [Background] Horacek TM, White AA, Greene GW, Reznar MM, Quick VM, Morrell JS, Colby SM, Kattelmann KK, Herrick MS, Shelnutt KP, Mathews A, Phillips BW, Byrd-Bredbenner C. Sneakers and spokes: an assessment of the walkability and bikeability of U.S. postsecondary institutions. J Environ Health. 2012 Mar;74(7):8-15; quiz 42. PMID 22428317
- [Background] O'Toole TP, Aaron KF, Chin MH, Horowitz C, Tyson F. Community-based participatory research: opportunities, challenges, and the need for a common language. J Gen Intern Med. 2003 Jul;18(7):592-4. doi: 10.1046/j.1525-1497.2003.30416.x. No abstract available. PMID 12848844
- [Background] Schultz JT, Moodie M, Mavoa H, Utter J, Snowdon W, McCabe MP, Millar L, Kremer P, Swinburn BA. Experiences and challenges in implementing complex community-based research project: the Pacific Obesity Prevention in Communities project. Obes Rev. 2011 Nov;12 Suppl 2:12-9. doi: 10.1111/j.1467-789X.2011.00911.x. PMID 22008555
- [Background] Szymona K, Quick V, Olfert M, et al. The University Environment: A Comprehensive Assessment of Health-Related Advertisements. Health Ed. 2012;112(6):497-512.
- [Derived] El Zein A, Colby SE, Zhou W, Shelnutt KP, Greene GW, Horacek TM, Olfert MD, Mathews AE. Food Insecurity Is Associated with Increased Risk of Obesity in US College Students. Curr Dev Nutr. 2020 Jul 15;4(8):nzaa120. doi: 10.1093/cdn/nzaa120. eCollection 2020 Aug. PMID 32793850
- [Derived] Olfert MD, Barr ML, Mathews AE, Horacek TM, Riggsbee K, Zhou W, Colby SE. Life of a vegetarian college student: Health, lifestyle, and environmental perceptions. J Am Coll Health. 2022 Jan;70(1):232-239. doi: 10.1080/07448481.2020.1740231. Epub 2020 Apr 28. PMID 32343196
- [Derived] El Zein A, Shelnutt KP, Colby S, Vilaro MJ, Zhou W, Greene G, Olfert MD, Riggsbee K, Morrell JS, Mathews AE. Prevalence and correlates of food insecurity among U.S. college students: a multi-institutional study. BMC Public Health. 2019 May 29;19(1):660. doi: 10.1186/s12889-019-6943-6. PMID 31142305
- [Derived] Famodu OA, Barr ML, Holaskova I, Zhou W, Morrell JS, Colby SE, Olfert MD. Shortening of the Pittsburgh Sleep Quality Index Survey Using Factor Analysis. Sleep Disord. 2018 Apr 12;2018:9643937. doi: 10.1155/2018/9643937. eCollection 2018. PMID 29850262
- [Derived] Loso J, Staub D, Colby SE, Olfert MD, Kattelmann K, Vilaro M, Colee J, Zhou W, Franzen-Castle L, Mathews AE. Gardening Experience Is Associated with Increased Fruit and Vegetable Intake among First-Year College Students: A Cross-Sectional Examination. J Acad Nutr Diet. 2018 Feb;118(2):275-283. doi: 10.1016/j.jand.2017.09.005. Epub 2017 Dec 1. PMID 29198845
- See also: Click here for more information about "Get Fruved": A Peer-Led, Train-the-Trainer Social Marketing Intervention to Increase Fruit and Vegetable Intake and Prevent Childhood Obesity A USDA grant-funded project — http://fruved.com/